CLINICAL TRIAL: NCT03443063
Title: An Open-label, Parallel-Group Study to Evaluate the Pharmacokinetics of Lemborexant and Its Metabolites in Subjects With Normal Renal Function or With Severe Renal Impairment
Brief Title: Study to Evaluate the Pharmacokinetics of Lemborexant (E2006) and Its Metabolites in Subjects With Normal Renal Function or With Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2006-A001-105
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2018-07

CONDITIONS: Renal Impairment
Keywords: severe renal impairment; lemborexant; normal renal function; healthy participants; metabolites; E2006; pharmacokinetics
MeSH Terms: conditions — Renal Insufficiency | interventions — lemborexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Severe Renal Impairment (Experimental): Participants with severe renal impairment (estimated glomerular filtration rate [eGFR] 15 to 29 milliliters per minute (mL/min/1.73 square meter [m^2]) and not on dialysis) will receive a single dose of 10 milligrams (mg) lemborexant (oral tablet) in the morning after an overnight fast.
  Interventions: Drug: Lemborexant
- Group 2: Normal Renal Function (Experimental): Participants with normal renal function (eGFR ≥90 mL/min/1.73 m^2) demographically matched to participants in Group 1 will receive a single dose of 10 mg lemborexant (oral tablet) in the morning after an overnight fast.
  Interventions: Drug: Lemborexant

INTERVENTIONS:
Drug: Lemborexant — oral tablet
  Other Names: E2006

SUMMARY:
This study will be conducted to assess the effect of severe renal impairment on the pharmacokinetics of lemborexant after a single-dose administration.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for All Participants:

* Male or female participants, ages 18 to 79 years, inclusive, at the time of informed consent.
* Body Mass Index between 18 and 40 kilograms per meters squared (kg/m^2), inclusive, at Screening.
* Voluntary agreement to provide written informed consent, and the willingness and ability to comply with all aspects of the protocol.
* Nonsmokers or smokers who smoke 20 cigarettes or less per day.
* Participants with normal liver function.

Additional Inclusion Criteria for Healthy Participants:

* Estimated glomerular filtration rate (eGFR) is ≥ 90 mL/min/1.73 m^2, as determined by the Modification of Diet in Renal Disease (MDRD) formula.

Additional Inclusion Criteria for Participants with Renal Impairment:

- Diagnosis of severe renal impairment (eGFR is 15 to 29 mL/min/1.73 m^2, as determined by the MDRD formula) that has been stable (without any change in disease status) for 60 days prior to study Screening and is confirmed on Day -1, as determined by the investigator by MDRD formula. If the renal function classification for the participant changed from screening to Day -1, eGFR should be repeated once within 24 to 48 hours. If eGFR variability across these scheduled and repeat time points indicates the participant does not consistently meet the criteria for one renal category group, participant enrollment into a renal category group will be at the discretion of the medical monitor and investigator, in consultation with the Sponsor.

Exclusion Criteria:

Exclusion Criteria for All Participants:

* Females who are breastfeeding or pregnant at Screening or Baseline.
* Females of childbearing potential who did not use a highly effective method of contraception within 28 days before study entry, or who did not agree to use an approved method of contraception from 28 days before study entry, throughout the entire study period, and for 28 days after study drug discontinuation.
* Intake of food supplements (including herbal preparations), foods or beverages that may affect cytochrome P450 (CYP) 3A4 (CYP3A4) enzyme (e.g., alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [e.g., kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard] and charbroiled meats) within 2 weeks before dosing until study discharge.
* Use of an herbal preparation containing Saint John's Wort within 4 weeks before dosing until study discharge.
* Known to be positive for human immunodeficiency virus.
* Presence of acute and active liver disease, or acute liver injury, as indicated by (1) an abnormal liver function test, or (2) clinical or laboratory signs of acute, active viral hepatitis (including B and C as demonstrated by positive serology at Screening). Participants with stable, chronic, inactive viral hepatitis B or C may be enrolled based on investigator's opinion.
* Corrected QT interval for heart rate on electrocardiograms (ECGs) by Fridericia's formula (QTcF) >480 milliseconds (msec) at Screening or Day -1. Before excluding a participant with QTcF >480 msec at Screening, ECG should be repeated once to confirm.
* A known or suspected history of drug or alcohol abuse disorder within 6 months prior to Screening.
* A positive urine drug test or a positive breathalyzer alcohol test at Screening or Day -1.
* Participation in another interventional clinical trial within 4 weeks, or 5 times the half-life of the investigational drug (whichever is longer), of lemborexant administration.
* Engaged in heavy/strenuous physical exercise within 2 weeks prior to check-in on Day -1 (e.g., marathon runners, weight lifters).
* Unwilling to abide by the study requirements, or in the opinion of the investigator, is not likely to complete the study.
* History of clinically significant drug or food allergies, or is presently experiencing significant seasonal allergies.
* Recent weight change that is considered clinically significant by the Investigator.
* Clinically significant findings revealed by physical examination, assessment of vital signs, ECG, or clinical laboratory testing.
* Use of any prohibited prescription or over-the-counter medication within 2 weeks or 5 half-lives (whichever is longer) before Screening, or plans to use any such treatment during the study. For participants with renal impairment, chronic stable administration of medications necessary for maintaining the clinical status of the participant may be permitted after consultation with the Medical Monitor.

Additional Exclusion Criteria for Healthy Participants:

* Presence of clinically significant illness requiring treatment or that may influence the outcome of the study (e.g., psychiatric disorders, disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system), a history of myocardial infraction, or a congenital abnormality.
* Receipt or donation of blood or blood products within 4 to 8 weeks prior to study drug administration.

Additional Exclusion Criteria for Participants With Renal Impairment:

* Any history of renal transplant.
* Any known significant bleeding diathesis (e.g., history of recent bleeding from esophageal varices), which could preclude multiple venipuncture or deep intramuscular injections.
* New significant illness that onset within 2 weeks prior to study drug administration.
* Current clinically relevant disease other than the renal impairment (e.g., cardiac, hepatic, gastrointestinal disorder, or a condition which may impact drug absorption), as determined by the investigator. Participants with a history of Type I or Type II diabetes may be eligible, providing that, in the investigator's opinion, the disease has been stable. Participants receiving insulin therapy may be eligible provided they have been on a stable (i.e., dose has not changed) treatment for at least 2 weeks prior to study enrollment and will continue the treatment throughout the study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United states from 07 February 2018 to 24 August 2018.
Pre-assignment Details: A total of 48 participants were screened, of which 32 were screen failures and 16 were enrolled and received study treatment.
Groups:
- Lemborexant: Severe Renal Impairment: Participants with severe renal impairment (estimated glomerular filtration rate [eGFR] 15 to 29 milliliters per minute (mL/min/1.73 square meter [m^2]) and not on dialysis) received a single dose of 10 milligrams (mg) lemborexant (oral tablet) on Day 1 in the morning after an overnight fast.
- Lemborexant: Normal Renal Function: Participants with normal renal function (eGFR greater than or equal to (>=) 90 mL/min/1.73 m^2) demographically matched to participants with severe renal impairment (matched according to age, race, sex, and body mass index [BMI]) received a single dose of 10 mg lemborexant (oral tablet) on Day 1 in the morning after an overnight fast.
Period: Overall Study
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set was the group of participants who were dosed with the test drug and had at least one postdose safety assessment.
Groups:
- Lemborexant: Severe Renal Impairment: Participants with severe renal impairment (eGFR 15 to 29 mL/min/1.73 m^2 and not on dialysis) received a single dose of 10 mg lemborexant (oral tablet) on Day 1 in the morning after an overnight fast.
- Lemborexant: Normal Renal Function: Participants with normal renal function (eGFR >=90 mL/min/1.73 m^2) matched to participants with severe renal impairment (matched according to age, race, sex, and BMI) received a single dose of 10 mg lemborexant (oral tablet) on Day 1 in the morning after an overnight fast.
- Total: Total of all reporting groups
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (5.40) | 66.5 (7.91) | 66.9 (6.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Lemborexant
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: The pharmacokinetic (PK) analysis set was the group of participants who were dosed with the test drug and had sufficient PK data to derive at least one PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Lemborexant: Normal Renal Function: Participants with normal renal function (eGFR >=90 mL/min/1.73 m^2) demographically matched to participants with severe renal impairment (matched according to age, race, sex, and BMI) received a single dose of 10 mg lemborexant (oral tablet) on Day 1 in the morning after an overnight fast.
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
nanogram per milliliter (ng/mL) | 48.9 (41.0) | 46.6 (29.2)
Statistical Analysis 1: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Test type: Other; Percent (%) ratio of geometric means = 104.83, 90% CI 2-sided [77.41 to 141.97] — Percent ratio was calculated by dividing the geometric mean of reporting arm "Lemborexant: Severe Renal Impairment" by geometric mean of reporting arm "Lemborexant: Normal Renal Function", then multiplying the value by 100

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 72 Hours Post Dose (AUC[0-72h]) of Lemborexant
Time Frame: Day 1: predose, 0.5 up to 72 hours postdose
Population: The PK analysis set was the group of participants who were dosed with the test drug and had sufficient PK data to derive at least one PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
hour*nanogram per milliliter (h*ng/mL) | 419 (21.9) | 315 (27.4)
Statistical Analysis 1: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Test type: Other; Percent (%) ratio of geometric means = 133.03, 90% CI 2-sided [107.30 to 164.93] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC[0-t]) of Lemborexant
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
h*ng/mL | 660 (29.3) | 439 (36.9)
Statistical Analysis 1: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Test type: Other; Percent (%) ratio of geometric means = 150.53, 90% CI 2-sided [113.16 to 200.26] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUC[0-inf]) of Lemborexant
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: The PK analysis set was the group of participants who were dosed with the test drug and had sufficient PK data to derive at least one PK parameter. Here "overall number of participants analyzed" signifies the participants who were evaluable for analysis for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 7 | 7
h*ng/mL | 672 (19.6) | 449 (38.3)
Statistical Analysis 1: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Test type: Other; Percent (%) ratio of geometric means = 149.84, 90% CI 2-sided [113.06 to 198.58] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Metabolites of Lemborexant (M4, M9, and M10)
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
ng/mL
  Metabolite M4 | 6.37 (44.8) | 7.96 (39.5)
  Metabolite M9 | 3.77 (44.1) | 4.74 (45.9)
  Metabolite M10 | 2.78 (50.5) | 3.83 (48.0)
Statistical Analysis 1: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M4; Test type: Other; Percent (%) ratio of geometric means = 80.09, 90% CI 2-sided [56.07 to 114.40] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M9; Test type: Other; Percent (%) ratio of geometric means = 79.51, 90% CI 2-sided [54.48 to 116.03] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M10; Test type: Other; Percent (%) ratio of geometric means = 72.49, 90% CI 2-sided [48.08 to 109.29] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Lemborexant and Its Metabolites (M4, M9, and M10)
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: as for outcome 2
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
hour (h)
  Lemborexant | 1.00 [0.50 to 3.00] | 1.00 [1.00 to 1.50]
  Metabolite M4 | 3.50 [1.00 to 4.00] | 2.00 [1.00 to 4.00]
  Metabolite M9 | 1.00 [1.00 to 4.00] | 1.25 [1.00 to 2.00]
  Metabolite M10 | 5.00 [3.00 to 72.17] | 3.00 [2.00 to 4.00]

7. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 8 Hours Post Dose (AUC[0-8h]) of Lemborexant and Its Metabolites (M4, M9, and M10)
Time Frame: Day 1: predose, 0.5 up to 8 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
h*ng/mL
  Lemborexant | 159 (23.2) | 143 (21.2)
  Metabolite M4 | 36.9 (46.2) | 45.9 (34.9)
  Metabolite M9 | 16.7 (31.8) | 19.2 (35.7)
  Metabolite M10 | 15.9 (63.8) | 24.4 (49.1)
Statistical Analysis 1: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Lemborexant; Test type: Other; Percent (%) ratio of geometric mean = 111.25, 90% CI 2-sided [91.69 to 134.99] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M4; Test type: Other; Percent (%) ratio of geometric means = 80.28, 90% CI 2-sided [56.81 to 113.46] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M9; Test type: Other; Percent (%) ratio of geometric means = 86.71, 90% CI 2-sided [64.92 to 115.81] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M10; Test type: Other; Percent (%) ratio of geometric means = 65.38, 90% CI 2-sided [41.08 to 104.04] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 72 Hours Post Dose (AUC[0-72h]) of Metabolites of Lemborexant (M4, M9, and M10)
Time Frame: Day 1: predose, 0.5 up to 72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
h*ng/mL
  Metabolite M4 | 164 (19.0) | 143 (25.3)
  Metabolite M9 | 67.2 (16.8) | 53.8 (31.9)
  Metabolite M10 | 149 (40.2) | 162 (34.7)
Statistical Analysis 1: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M4; Test type: Other; Percent (%) ratio of geometric means = 114.69, 90% CI 2-sided [94.45 to 139.28] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M9; Test type: Other; Percent (%) ratio of geometric means = 124.94, 90% CI 2-sided [100.27 to 155.67] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M10; Test type: Other; Percent (%) ratio of geometric means = 92.05, 90% CI 2-sided [66.87 to 126.71] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC[0-t]) of Metabolites of Lemborexant (M4, M9, and M10)
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
h*ng/mL
  Metabolite M4 | 247 (25.9) | 181 (32.9)
  Metabolite M9 | 106 (27.0) | 68.7 (35.8)
  Metabolite M10 | 322 (28.3) | 272 (40.9)
Statistical Analysis 1: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M4; Test type: Other; Percent (%) ratio of geometric means = 136.28, 90% CI 2-sided [105.62 to 175.85] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M9; Test type: Other; Percent (%) ratio of geometric means = 154.29, 90% CI 2-sided [117.53 to 202.57] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M10; Test type: Other; Percent (%) ratio of geometric means = 118.54, 90% CI 2-sided [87.84 to 159.97] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Area Under the Plasma Concentration-Time Curve Extrapolated to Infinity (AUC[0-inf]) of Metabolites of Lemborexant (M4, M9, and M10)
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: The PK analysis set was the group of participants who were dosed with the test drug and had sufficient PK data to derive at least one PK parameter. Here "number analyzed" signifies the participants who were evaluable for analysis for specific metabolite of lemborexant for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
h*ng/mL
  Metabolite M4: number analyzed (Participants) | 7 | 7
  Metabolite M4 | 248 (20.4) | 179 (29.9)
  Metabolite M9: number analyzed (Participants) | 7 | 7
  Metabolite M9 | 108 (24.1) | 73.5 (38.8)
  Metabolite M10: number analyzed (Participants) | 5 | 6
  Metabolite M10 | 357 (20.1) | 262 (36.7)
Statistical Analysis 1: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M4; Test type: Other; Percent (%) ratio of geometric means = 138.62, 90% CI 2-sided [109.10 to 176.14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M9; Test type: Other; Percent (%) ratio of geometric means = 147.03, 90% CI 2-sided [109.06 to 198.22] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M10; Test type: Other; Percent (%) ratio of geometric means = 136.42, 90% CI 2-sided [98.19 to 189.54] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Area Under the Plasma Concentration-Time Curve Adjusted by Unbound Fraction of Plasma (AUCu) of Lemborexant and Its Metabolites (M4, M9, and M10)
Description: AUCu was defined as the AUC(0-inf) adjusted by unbound fraction in plasma, and calculated by multiplying the value of AUC(0-inf) with Plasma protein unbound fraction (fu).
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: The PK analysis set was the group of participants who were dosed with the test drug and had sufficient PK data to derive at least one PK parameter. Here "number analyzed" signifies the participants who were evaluable for analysis for lemborexant and for specific metabolite of lemborexant for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
h*ng/mL
  Lemborexant: number analyzed (Participants) | 7 | 7
  Lemborexant | 45.7 (16.9) | 32.4 (44.3)
  Metabolite M4: number analyzed (Participants) | 6 | 7
  Metabolite M4 | 57.8 (12.6) | 46.4 (27.0)
  Metabolite M9: number analyzed (Participants) | 6 | 7
  Metabolite M9 | 16.6 (13.3) | 11.6 (38.0)
  Metabolite M10: number analyzed (Participants) | 5 | 6
  Metabolite M10 | 32.1 (28.2) | 22.9 (36.5)
Statistical Analysis 1: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Lemborexant; Test type: Other; Percent (%) ratio of geometric means = 141.07, 90% CI 2-sided [103.79 to 191.73] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M4; Test type: Other; Percent (%) ratio of geometric means = 124.48, 90% CI 2-sided [100.58 to 154.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M9; Test type: Other; Percent (%) ratio of geometric means = 143.31, 90% CI 2-sided [107.72 to 190.65] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Lemborexant: Severe Renal Impairment vs Lemborexant: Normal Renal Function; Metabolite M10; Test type: Other; Percent (%) ratio of geometric means = 140.20, 90% CI 2-sided [98.11 to 200.35] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Percentage of AUC(0-inf) Based on Extrapolation (AUCex) of Lemborexant and Its Metabolites (M4, M9, and M10)
Description: AUCex was calculated by dividing the difference of (AUC(0-inf) and AUC(0-t)) by value of AUC(0-inf) and then multiplying the value by 100.
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUCex
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
percentage of AUCex
  Lemborexant: number analyzed (Participants) | 7 | 7
  Lemborexant | 7.65 (73.1) | 5.74 (85.7)
  Metabolite M4: number analyzed (Participants) | 7 | 7
  Metabolite M4 | 5.35 (75.2) | 4.88 (24.6)
  Metabolite M9: number analyzed (Participants) | 7 | 7
  Metabolite M9 | 6.72 (69.0) | 6.15 (30.3)
  Metabolite M10: number analyzed (Participants) | 5 | 6
  Metabolite M10 | 7.46 (79.5) | 7.16 (74.1)

13. Secondary Outcome: Observed Terminal Elimination Half-life (t1/2) of Lemborexant and Its Metabolites (M4, M9, and M10)
Description: Terminal plasma half-life is the time required for plasma/blood concentration to decrease by 50%. This is not the time required to eliminate half the administered dose.
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: as for outcome 11
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
hour (h)
  Lemborexant: number analyzed (Participants) | 7 | 7
  Lemborexant | 79.5 [52.3 to 93.4] | 79.7 [44.8 to 86.5]
  Metabolite M4: number analyzed (Participants) | 7 | 7
  Metabolite M4 | 68.1 [47.5 to 83.1] | 67.0 [38.1 to 82.8]
  Metabolite M9: number analyzed (Participants) | 7 | 7
  Metabolite M9 | 64.1 [43.0 to 96.9] | 53.5 [27.6 to 81.0]
  Metabolite M10: number analyzed (Participants) | 5 | 6
  Metabolite M10 | 63.4 [43.1 to 93.5] | 70.5 [29.4 to 84.2]

14. Secondary Outcome: Observed Elimination Rate Constant (LambdaZ) of Lemborexant and Its Metabolites (M4, M9, and M10)
Description: Estimated by linear regression through at least three data points (not including tmax) in the terminal phase of the log concentration-time profile.
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: per hour (1/h)
Groups:
- Lemborexant: Normal Renal Function: Participants with normal renal function (eGFR >=90 mL/min/1.73 m^2) demographically matched to participants with severe renal impairment (matched according to age, race, sex, and BMI) received a single dose of 10 mg lemborexant (oral tablet) in the morning on Day 1 after an overnight fast.
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
per hour (1/h)
  Lemborexant: number analyzed (Participants) | 7 | 7
  Lemborexant | 0.00950 (25.4) | 0.0102 (28.7)
  Metabolite M4: number analyzed (Participants) | 7 | 7
  Metabolite M4 | 0.0108 (21.5) | 0.0114 (30.2)
  Metabolite M9: number analyzed (Participants) | 7 | 7
  Metabolite M9 | 0.0113 (29.7) | 0.0142 (47.8)
  Metabolite M10: number analyzed (Participants) | 5 | 6
  Metabolite M10 | 0.0111 (30.5) | 0.0114 (39.2)

15. Secondary Outcome: Apparent Body Clearance (CL/F) of Lemborexant
Description: CL/F is the clearance for parent Lemborexant only and was calculated as Dose/[AUC0-inf]. Blood samples were analyzed for the amount of Lemborexant in the plasma.
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 7 | 7
liter per hour (L/h) | 14.9 (19.6) | 22.3 (38.3)

16. Secondary Outcome: Apparent Volume of Distribution (Vz/F) Based on the Terminal Phase of Lemborexant
Description: The apparent volume of distribution gives information about the amount of Lemborexant distributed in body tissue rather than the blood/plasma. Vz/F for parent Lemborexant only was calculated as Dose /([ λz]*[AUC0-inf]).
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter (L)
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 7 | 7
liter (L) | 1570 (32.8) | 2180 (46.3)

17. Secondary Outcome: Metabolite-to-Parent Ratio of AUC(0-inf), Corrected for Molecular Weights (MPR AUC[0-inf]) of Metabolites of Lemborexant (M4, M9, and M10)
Description: The AUC metabolite to parent ratio (MPR) is the ratio of AUC(0-inf) of the individual metabolite to AUC(0-inf) of lemborexant, corrected for molecular weights.
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
ratio
  Metabolite M4: number analyzed (Participants) | 7 | 7
  Metabolite M4 | 0.355 (7.49) | 0.384 (13.6)
  Metabolite M9: number analyzed (Participants) | 7 | 6
  Metabolite M9 | 0.155 (18.5) | 0.150 (31.7)
  Metabolite M10: number analyzed (Participants) | 5 | 6
  Metabolite M10 | 0.549 (13.4) | 0.612 (10.3)

18. Secondary Outcome: Plasma Protein Unbound Fraction (Fu) of Lemborexant and Its Metabolites (M4, M9, and M10)
Description: Unbound fraction of drug in plasma was calculated as 100% minus (-) mean percent of Lemborexant and Its Metabolites M4. M9. M10 bound to plasma protein for each participant.
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: % unbound
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
% unbound
  Lemborexant | 6.68 (10.4) | 7.11 (10.7)
  Metabolite M4: number analyzed (Participants) | 7 | 8
  Metabolite M4 | 24.1 (11.4) | 25.5 (6.90)
  Metabolite M9: number analyzed (Participants) | 7 | 8
  Metabolite M9 | 15.7 (12.5) | 16.1 (8.79)
  Metabolite M10: number analyzed (Participants) | 7 | 8
  Metabolite M10 | 8.18 (27.5) | 8.63 (11.9)

19. Secondary Outcome: Apparent Clearance Relative to the Unbound Plasma Concentration (CLu/F) Based on AUCu of Lemborexant
Description: Unbound fraction of drug in plasma was calculated as 100% - mean percent of Lemborexant bound to plasma protein for each participant.
Time Frame: Day 1: predose, 0.5 up to 240 hours postdose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/h)
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 7 | 7
liter per hour (L/h) | 219 (16.9) | 309 (44.3)

20. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Up to Day 11
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
Participants
  TEAEs | 5 | 7
  SAEs | 0 | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Time Frame: Up to Day 11
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

22. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Vital Sign Values
Time Frame: Up to Day 11
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

23. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Parameter Values
Time Frame: Up to Day 11
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Lemborexant: Severe Renal Impairment: Participants with severe renal impairment (eGFR 15 to 29 mL/min/1.73 m^2 and not on dialysis) received a single dose of 10 mg lemborexant (oral tablet) in the morning after an overnight fast.
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 11
Description: AEs were collected for the participants who were in the safety analysis set (all participants who were dosed with the test drug and had at least one postdose safety assessment).
Arm/Group | Lemborexant: Severe Renal Impairment | Lemborexant: Normal Renal Function
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 5/8 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lemborexant: Severe Renal Impairment (N=8) | Lemborexant: Normal Renal Function (N=8)
Chills (General disorders) | 1 | 0
Somnolence (Nervous system disorders) | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/63/NCT03443063/Prot_002.pdf
  • Statistical Analysis Plan (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/63/NCT03443063/SAP_004.pdf